CLINICAL TRIAL: NCT06499870
Title: Optimizing Treatment and Advanced Multi-Imaging Response Evaluation for Very-High-Risk Prostate Cancer (OPTIMAL) - a Phase II Single Arm Study
Brief Title: Relugolix and Enzalutamide in Combination With Radiation Therapy for the Treatment of Very High Risk Prostate Cancer, OPTIMAL Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 24U02; NCI-2024-03934 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00221219; NU 24U02 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — Biopsy; Specimen Handling; enzalutamide; 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid; Radiotherapy, Image-Guided; Magnetic Resonance Spectroscopy; relugolix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (relugolix, enzalutamide, IGRT) (Experimental): Patients receive relugolix PO QD and enzalutamide PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 18 months in the absence of disease progression or unacceptable toxicity. After 4 months of treatment with relugolix and enzalutamide, patients begin IGRT per standard of care. Patients also undergo fluorine F 18 piflufolastat PET/MRI and CT on the trial, undergo collection of blood samples throughout the trial, and undergo biopsy during follow up.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Enzalutamide; Other: Fluorine F 18 Piflufolastat; Radiation: Image Guided Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Relugolix

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV 3100; MDV-3100; MDV3100; Xtandi
Other: Fluorine F 18 Piflufolastat — Undergo fluorine F 18 piflufolastat PET/MRI
  Other Names: 18F-DCFPyL; Fluorine F 18 DCFPyL; Piflufolastat F 18; Piflufolastat F-18; Piflufolastat F18; Pylarify
Radiation: Image Guided Radiation Therapy — Undergo IGRT
  Other Names: IGRT; image-guided radiation therapy; Image-Guided Radiotherapy
Procedure: Magnetic Resonance Imaging — Undergo PET/MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Questionnaire Administration — Ancillary studies
Drug: Relugolix — Given PO
  Other Names: N-(4-(1-((2,6-Difluorophenyl)methyl)-5-((dimethylamino)methyl)-1,2,3,4-tetrahydro-3-(6-methoxy-3-pyridazinyl)-2,4-dioxothieno(2,3-d)pyrimidin-6-yl)phenyl)-N'-methoxyurea; Orgovyx; Relumina; TAK 385; TAK-385; TAK385

SUMMARY:
This phase II trial tests how well relugolix and enzalutamide, in combination with radiation therapy, works in treating patients with very high risk prostate cancer. Relugolix is a form of androgen deprivation therapy. It prevents the release of testosterone, a hormone required to sustain prostate growth. Reducing testosterone levels may inhibit the proliferation of prostate tumor cells that need testosterone to grow. Enzalutamide is an androgen receptor signaling inhibitor. It inhibits the activity of prostate tumor cell receptors, which may reduce proliferation of prostate tumor cells. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. Adding relugolix and enzalutamide to radiation therapy may be more effective at treating patients with very high risk prostate cancer than giving any of these treatments alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy of radiation therapy (RT) with androgen deprivation therapy (ADT) (relugolix) and an androgen receptor signaling inhibitor (enzalutamide), for a total duration of 18 months, in patients with National Comprehensive Cancer Network (NCCN) very high-risk prostate cancer, as determined by a 2-year biopsy positivity rate.

SECONDARY OBJECTIVES:

I. To determine the 4-year disease free survival (DFS) (biochemical failure of prostate specific antigen [PSA] nadir +2ng/mL, local or regional recurrence, distant metastasis, or death from any cause).

II. To evaluate testosterone recovery.

EXPLORATORY OBJECTIVES:

I. To evaluate impact on patient-reported health-related quality of life utilizing (1) Expanded Prostate Cancer Index Composite, EPIC-26 and (2) European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLC-C30).

II. To investigate a relationship between magnetic resonance imaging (MRI)-positron emission tomography (PET) radiomic response (baseline and after neoadjuvant therapy) correlated with pathologic and disease control endpoints.

OUTLINE:

Patients receive relugolix orally (PO) once daily (QD) and enzalutamide PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 18 months in the absence of disease progression or unacceptable toxicity. After 4 months of treatment with relugolix and enzalutamide, patients begin image-guided radiation therapy (IGRT) per standard of care. Patients also undergo fluorine F 18 piflufolastat PET/MRI and CT on the trial, undergo collection of blood samples throughout the trial, and undergo biopsy during follow up.

After completion of study treatment, patients are followed up every 3-6 months for up to 30 months (48 months after study registration).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed prostate adenocarcinoma consistent with NCCN very-high-risk (VHR) prostate cancer defined with at least one of the following:

  * cT3b-cT4 (American Joint Committee on Cancer [AJCC] 9.0)
  * > 4 cores with grade group 4 or 5 prostate cancer
  * Primary gleason pattern 5
  * 2 or 3 NCCN high-risk features.
* Patients with involved pelvic lymph nodes below the common iliac bifurcation will be allowed as long as the criteria for VHR (very-high risk) are met
* Patients must be age ≥ 18 years
* Patients must have testosterone > 50 ng/dL within 90 days prior to registration

  * Note: Prior androgen deprivation (gonadotrophin releasing hormone [GnRH] analog and/or non-steroidal antiandrogen) therapy is allowed provided that it is less than 60 days of prior total duration and that serum testosterone concentration must be ≥ 50 ng/dL prior to enrollment; 5-alpha reductase inhibitors will not impact eligibility, but must be discontinued prior to starting protocol treatment
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Leukocytes (white blood cells [WBC]) ≥ 2,500/mcL
* Absolute neutrophil count (ANC) ≥ 1,500/mcL
* Hemoglobin (Hgb) ≥ 8 g/dL
* Platelets (PLT) ≥ 80,000/mcL
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) ≤ 3 x institutional upper limit of normal (ULN)
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 3 x institutional ULN
* Creatinine ≤ institutional ULN
* Glomerular filtration rate (GFR) ≥ 30 mL/min/1.73 m^2

  * Estimated GFR (eGFR) is estimated GFR calculated by the abbreviated Modification of Diet in Renal Disease (MDRD) equation
* For patients with a known history of human immunodeficiency virus (HIV), infected patients on effective anti-retroviral therapy must have a viral load undetectable for 3 months prior to registration with a CD4 count of ≥ 200 cells/μL. Note also that HIV testing is not required for eligibility for this protocol as it is self-reported
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be better than class III
* Patients must not have contraindications to magnetic resonance (MR) imaging and be able to lie flat and still for approximately 30-40 minutes and be able to tolerate PET/CT imaging and radiation therapy treatment planning and delivery
* Patients with female partners of reproductive potential must agree to use effective contraception during treatment with and for 3 months after the last dose. Male patients must use a condom during sex with a pregnant woman
* Patients must have the ability to understand and the willingness to sign a written informed consent document and comply with the study requirements

Exclusion Criteria:

* Patients with definitive clinical or radiologic evidence of metastatic disease
* Patients with prior invasive malignancy (except non-melanomatous skin cancer carcinoma in situ of the male breast, penis, oral cavity, or stage Ta of the bladder, or stage I completely resected melanoma) unless disease free for a minimum of 2 years
* Prior radiotherapy that would result in overlap of radiation therapy fields
* Patients who have a history of any of the following:

  * History of documented inflammatory bowel disease
  * Symptomatic congestive heart failure (New York Heart Association Functional Classification III/IV) within 4 months prior to registration
  * Unstable angina pectoris requiring hospitalization within the last 4 months prior to registration
  * History of seizure disorder or condition that may yield a high risk of seizure (e.g., prior cortical stroke or significant brain trauma)
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * History of repeated falls and fractures over the past 12 months that in the opinion of the treating investigator would put the patient at risk for poor bone outcomes from androgen receptor targeted therapy
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
  * Patients with the inability to take oral medication OR have malabsorption syndrome or any other uncontrolled gastrointestinal condition (eg, nausea, diarrhea, vomiting) that might impair the bioavailability of enzalutamide and relugolix

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2028-11-19 (Estimated); Study Completion 2032-11-19 (Estimated)

PRIMARY OUTCOMES:
Pathologic response (biopsy positivity rate) | At 2 years
  Will determine the efficacy of radiation therapy with relugolix and enzalutamide, for a total duration of 18 months, in patients with National Comprehensive Cancer Network very high-risk prostate cancer, by a 2-year biopsy positivity rate.

SECONDARY OUTCOMES:
Disease-free survival | Up to 4 years
  Will be determined by biochemical failure of prostate specific antigen nadir + 2ng/mL, local or regional recurrence, distant metastasis, or death. Median survival time will be estimated with corresponding 95% confidence intervals.
Testosterone recovery | Up to 4 years
  Testosterone recovery will be defined as a total serum testosterone of ≥ 200 ng/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Sachdev, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States